CLINICAL TRIAL: NCT06831578
Title: Analgesic Efficacy of Ultrasound-guided Serratus Anterior Plane Block Versus Thoracic Paravertebral Plane Block in Patients Undergoing Thoracotomy
Brief Title: Compare the Perioperative Analgesic Effect of Ultrasound Guided Thoracic Paravertebral Block and Ultrasound Guided Serratus Anterior Block in Patients Undergoing Thoracotomy
Acronym: thoracotomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Hamza Sedky, lectuer of anathesia,intensive care and pain, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/2024 ANESTH
Record Dates: First submitted 2025-02-09; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2024-05

CONDITIONS: Thoracotomy; Thoracotomy Analgesia
Keywords: analgesia; thoracotomy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Consenting patients will be assigned randomly (1:1) into two groups. Both groups will receive general anesthesia and after induction an ultrasound guided serratu anterior plan block will be performed for one group and an ultrasound guided paravertebral plan block will be performed for the other. In both groups a loading dose of the local anesthetic (LA) solution( 20 ml of 0.25% bupivacaine ) will be injected before the surgical procedure
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- serratus anterior plane block (Active Comparator)
  Interventions: Procedure: seratuse anterior plane block
- paravertebral plane block (Active Comparator)
  Interventions: Procedure: paravertebral plane block

INTERVENTIONS:
Procedure: seratuse anterior plane block — after patient consenting, induction of anathesia Under sterile conditions, and while the patients will be still on the lateral position with the diseased side up after induction of anesthesia, a linear ultrasound transducer (10-12 MHz) will be placed in a sagittal plane over the mid-clavicular region of the thoracic cage. Then counting down ribs till the seventh rib will be identified in the mid-axillar]y line. The following muscles will be identified overlying the sixth rib: the latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscle (deep and inferior). The needle (22-G, 50-mm Touhy needle) will be introduced in-plane with respect to the ultrasound probe targeting the plane deep to the serratus anterior muscle . Under continuous ultrasound guidance, 20 ml of 0.25% bupivacaine will be injected then a catheter will be threaded. A continuous infusion of 5 ml/hr of 0.125% bupivacaine will be then started through the catheter.
  Arms: serratus anterior plane block
Procedure: paravertebral plane block — after concenting patient, induction of anathesia Paravertebral plan block will be performed while the patient is still in lateral position and a linear ultrasound transducer (10-12 MHz) will be used for ultrasound guidance. A sagittal or transverse image can be obtained at the appropriate vertebral level. After image optimization, the Tuohy needle is advanced in plane until the tip rests in the thoracic paravertebral space. Injection of small amounts of fluid (hydrodissection) will aid in needle tip location. Saline or local anesthetic is injected through the Tuohy needle. The endpoint for a successful block is anterior displacement of the pleura. 20 ml of 0.25% bupivacaine will be injected then a catheter will be threaded. A continuous infusion of 5 ml/hr of 0.125% bupivacaine will be then started through the catheter. The catheter is threaded through the Tuohy needle and its position is confirmed by injecting local anesthetic or small air bubbles. Pleural depression should agai
  Arms: paravertebral plane block

SUMMARY:
The aim of this study is to compare the perioperative analgesic effect of ultrasound guided thoracic paravertebral block and ultrasound guided serratus anterior block in patients undergoing thoracotomy.

DETAILED DESCRIPTION:
randomized, comparative study General anesthesia will be conducted

ELIGIBILITY:
Inclusion Criteria:

* : Patients 20 to 60 years old
* ASA physical status of class II and III.

Exclusion Criteria:

Patients with severe respiratory disease

* preexisting neurologic deficit
* allergy to any of the study drug
* kypho-scoliosis
* presence of local infection
* on current chronic analgesic therapy, having history of opioid dependence'
* patient refusal
* inablity to communicate with the investigators
* who will require postoperative mechanical ventilation .

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
postoperative pain | postoperative up to 24 hours
  with the use of the visual analouge scale (VAS) in the preoperative visit. Where 0 score as no pain and 10 as the worst imaginable pain.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Menoufia university hospital, Shebeen Elkom, Menoufia
  - Menoufia faculty of medicine hospital, Shebin Elkom